CLINICAL TRIAL: NCT01006577
Title: Side-to-end Anastomosis Versus Colon J Pouch for Reconstruction After Low Anterior Resection for Rectal Cancer (SAVE)
Acronym: SAVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: ChirNet (Unknown)
Responsible Party: Dr. Johannes Lauscher; PD Dr. Jörg-Peter Ritz, Department of General, Vascular and Thoracic Surgery; Charité Campus Benjamin Franklin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EA4/105/08
Record Dates: First submitted 2009-10-19; First posted 2009-11-03 (Estimated); Last update posted 2009-11-03 (Estimated); Status verified 2009-11

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; side-to-end anastomosis; colon J pouch; fecal incontinence; anorectal function; Are there differences between side-to-end anastomosis and colon J pouch in; bowel function (fecal incontinence, frequency of bowel movements, rectal urgency, incomplete evacuation); quality of life; postoperative complications; operation time/ institutional costs
MeSH Terms: conditions — Rectal Neoplasms; Fecal Incontinence; Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- colon j pouch (Other): Control intervention: Low anterior resection for rectal cancer with total mesorectal excision (TME), ligation of the inferior mesenteric artery, mobilization of the splenic flexure, radical lymph node dissection and colon J pouch rectal/colon J pouch anal anastomosis (CJP). The colon J Pouch is formed by the descending colon by stapling. The intended minimal distal clearance margin from the tumor is 2 cm. A protective loop ileostomy will be performed regularly which is intended to be closed 3 months postoperatively.
  Interventions: Procedure: colon j pouch
- side-to-end anastomosis (STE) (Experimental): Experimental intervention: Low anterior resection for rectal cancer < 12 cm from the anal verge with total mesorectal excision (TME), ligation of the inferior mesenteric artery, mobilization of the splenic flexure, radical lymph node dissection and side-to-end colorectal/ coloanal anastomosis (STE). The blind end of the descending colon is closed with a linear stapler. The length of the blind end is measured and the integrity of the anastomosis is tested intraoperatively. The intended minimal distal clearance margin from the tumor is 2 cm. A protective loop ileostomy will be performed regularly which is intended to be closed 3 months postoperatively.
  Interventions: Procedure: side-to-end anastomosis

INTERVENTIONS:
Procedure: side-to-end anastomosis — Low anterior resection for rectal cancer < 12 cm from the anal verge with total mesorectal excision (TME), ligation of the inferior mesenteric artery close to the aorta, mobilization of the splenic flexure, radical lymph node dissection and side-to-end colorectal/ coloanal anastomosis (STE). The blind end of the descending colon (3-5 cm long) is closed with a linear stapler. Stapling of the anastomosis is done by introducing the stapler from the anus by the assistant surgeon while the surgeon is holding the descending colon in the correct position. The anastomosis is performed on the antimesenteric aspect of the descending colon. The length of the blind end is measured and the integrity of the anastomosis is tested intraoperatively. The intended minimal distal clearance margin from the tumor is 2 cm. A protective loop ileostomy will be performed regularly which is intended to be closed 3 months postoperatively.
  Arms: side-to-end anastomosis (STE)
Procedure: colon j pouch — Low anterior resection for rectal cancer with total mesorectal excision (TME), ligation of the inferior mesenteric artery close to the aorta, mobilization of the splenic flexure, radical lymph node dissection and colon J pouch rectal/colon J pouch anal anastomosis (CJP). The colon J Pouch is formed by the descending colon by stapling with a defined pouch limb length of 5-6 cm, which is measured intraoperatively. The stapling is done by introducing the stapler from the anus by the assistant surgeon while the surgeon is holding the descending colon in the correct position. The integrity of the anastomosis is tested intraoperatively. The intended minimal distal clearance margin from the tumor is 2 cm. A protective loop ileostomy will be performed regularly which is intended to be closed 3 months postoperatively.
  Arms: colon j pouch

SUMMARY:
Primary hypothesis: Side-to-end anastomosis is non-inferior to colon J pouch for reconstruction after low anterior resection for rectal cancer in fecal incontinence (Wexner score).

Research questions: Are there differences between side-to-end anastomosis and colon J pouch in

* bowel function (fecal incontinence, frequency of bowel movements, rectal urgency, incomplete evacuation)
* quality of life
* sexual function
* urinary function
* postoperative complications
* operation time/ institutional costs

DETAILED DESCRIPTION:
Experimental intervention: Low anterior resection for rectal cancer < 12 cm from the anal verge with total mesorectal excision (TME), ligation of the inferior mesenteric artery close to the aorta, mobilization of the splenic flexure, radical lymph node dissection and side-to-end colorectal/ coloanal anastomosis (STE). The blind end of the descending colon (3-5 cm long) is closed with a linear stapler. Stapling of the anastomosis is done by introducing the stapler from the anus by the assistant surgeon while the surgeon is holding the descending colon in the correct position. The anastomosis is performed on the antimesenteric aspect of the descending colon. The length of the blind end is measured and the integrity of the anastomosis is tested intraoperatively. The intended minimal distal clearance margin from the tumor is 2 cm. A protective loop ileostomy will be performed regularly which is intended to be closed 3 months postoperatively.

Control intervention: Low anterior resection for rectal cancer with total mesorectal excision (TME), ligation of the inferior mesenteric artery close to the aorta, mobilization of the splenic flexure, radical lymph node dissection and colon J pouch rectal/colon J pouch anal anastomosis (CJP). The colon J Pouch is formed by the descending colon by stapling with a defined pouch limb length of 5-6 cm, which is measured intraoperatively. The stapling is done by introducing the stapler from the anus by the assistant surgeon while the surgeon is holding the descending colon in the correct position. The integrity of the anastomosis is tested intraoperatively. The intended minimal distal clearance margin from the tumor is 2 cm. A protective loop ileostomy will be performed regularly which is intended to be closed 3 months postoperatively.

Follow-up per patient: 24 months postoperatively

ELIGIBILITY:
Inclusion Criteria:

* patients with histological proven middle to low rectal cancer (< 12 cm from the anal verge) requiring low anterior resection with TME
* with or without (neo)-adjuvant radiochemotherapy
* age ≥18 years
* normal preoperative sphincter status (Wexner score = 0)

Exclusion Criteria:

* synchronous metastasis
* age > 80 years
* previous colon resection
* inflammatory bowel disease
* previous pelvic malignant tumor
* no anterior resection/ TME possible
* synchronous other malignant disease
* emergency operation
* local excision by colonoscopy possible
* unability to complete or comprehend the preoperative questionnaire

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2010-06; Primary Completion 2015-07 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Side-to-end anastomosis is not inferior not colon J pouch in terms of fecal incontinence. fecal incontinence (Wexner score) | First patient in to last patient out: 03/2010 -03/2015

SECONDARY OUTCOMES:
anorectal function | 03/2010-03/2015
quality of life | 03/2010-03/2015
postoperative complications | 03/2010-03/2015
sexual function | 03/2010-03/2015
urinary function | 03/2010-03/2015
operation time | 03/2010-03/2015
institutional costs | 03/2010-03/2015
local recurrence | 03/2010-03/2015
cancer related deaths | 03/2010-03/2015

CONTACTS AND LOCATIONS:
Overall Officials: Johannes C Lauscher, MD, Principal Investigator — Charité Campus Benjamin Franklin; Department of General, Vascular and Thoracic Surgery; Jörg-Peter Ritz, PD Dr., Principal Investigator — Charité Campus Benjamin Franklin; Department of General, Vascular and Thoracic Surgery; Heinz J Buhr, Prof. Dr., Study Chair — Charité Campus Benjamin Franklin; Department of General, Vascular and Thoracic Surgery
Locations (1):
- Charité Campus Benjamin Franklin; Hindenburgdamm 30, Berlin, State of Berlin, Germany

REFERENCES:
- See also: Homepage of the Coordinating Center for Clinical Studies (Monitoring of the study) — http://www.kks.charite.de